CLINICAL TRIAL: NCT01761643
Title: CCTG 595: A Multicenter, Randomized Study of Text Messaging to Improve Adherence to PrEP in Risky MSM
Brief Title: CCTG 595: Text Messaging Intervention to Improve Adherence to PrEP in High-risk MSM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); City of Long Beach Department of Health and Human Services (Other Government); California HIV/AIDS Research Program (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTG 595
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Patient Adherence; HIV Seronegativity
Keywords: PrEP; Pre exposure Prophylaxis; Text Messaging; Truvada; iTab; CCTG; 595
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to evaluate a promising method of reinforcing PrEP adherence using text message. In this study, we will hope to learn if text message reminders increase PrEP adherence.
Masking Description: Group 1: PrEP daily, HIV/STI screening, adherence and risk behavior counseling, and safety monitoring Group 2: PrEP daily, HIV/STI screening, adherence and risk behavior counseling, and safety monitoring as well as iTAB text adherence reminders
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SoC) (No Intervention): This proposal will perform a study of potential methods to improve adherence and retention by evaluating standard procedures versus the use of the iTAB platform.
  All subjects will receive SoC that will include health education, clinical assessments, laboratory safety monitoring, STI and HIV screening, HIV risk reduction counseling, assessment of psycho-social barriers, adherence counseling, and completion of a computer based survey.
- SoC + iTab (Active Comparator): Subjects assigned to the iTAB intervention will receive daily dosing reminders that will be sent for the first 6 weeks and then continue with reminders for the duration of the study.
  Subjects will have visits with the study coordinator to introduce the iTAB texting system.
  Once the time is identified, the text reminder system is automated. Patients will confirm medication taking via text responses to the personalized reminders. If a participant does not respond on three consecutive occasions, a high alert message (chosen by the participant) will be sent. If the subject does not respond to this message, the study coordinator would initiate phone calls to contact the subject and explore barriers.
  Interventions: Device: SoC + iTab

INTERVENTIONS:
Device: SoC + iTab — Text messaging reminders to improve adherence to PrEP
  Arms: SoC + iTab

SUMMARY:
CCTG 595 is a controlled, open-label, two-arm, randomized (1:1) clinical demonstration project to determine if the use of a text-message based adherence intervention (iTAB) improves retention and adherence to PrEP compared to standard of care (SoC) PrEP delivery.

DETAILED DESCRIPTION:
A total of 400 HIV-uninfected men who have sex with men (MSM)and male to female (M to F) transgender individuals with recent high-risk transmission behavior will be enrolled into the study. Each subject will be followed for up to 48 weeks after enrollment of the last subject. The primary endpoint will be measured at 48 weeks.

All subjects will start PrEP with TDF + FTC fixed dose combination given once daily. Subjects will be randomized (1:1) to either the iTAB text messaging adherence reminder intervention with SoC or the SoC alone arm. Subjects placed into the iTAB intervention arm will receive a personalized, automated texting system to maintain adherence and retention. Both groups will receive access to PrEP in accordance with standardized comprehensive methods of prescribing, risk reduction counseling, adherence counseling, and clinical assessments that include safety monitoring, as well as HIV and STD screening.

TDF 300 mg + FTC 200 mg fixed dose combination will be given orally once daily starting at the baseline visit (month 0) and continued throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Man or transgender M to F who has sex with men.
* Age 18 years or older.
* Subjects must have substantial ongoing risk of acquisition of HIV as evident by one or more of the following:

  * Has at least one HIV infected sexual partner for ≥4 weeks.
  * No condom use during anal intercourse with ≥3 male sex partners who are HIV-positive or of unknown HIV status during the last 3 months.
  * No condom use during anal sex with ≥1 male partner and STI diagnosis during the last 3 months.
* Negative for HIV infection by rapid HIV test and confirmed negative by NAT or other sensitive method such as antibody- antigen test.
* Acceptable laboratory values in the past 30 days:

  * Calculated creatinine clearance of at least 60 mL/min by the Cockcroft-Gault formula (eCcr (male) in mL/min = [(140 - age in years) x (lean body weight in kg)] / (72 x serum creatinine in mg/dL)
  * Alanine aminotransferase (ALT) and/ or aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN)
  * Hemoglobin > 9 g/dL
  * Absolute neutrophil count > 750/ mm3
  * Platelets > 75,000/ mm3

Exclusion Criteria:

* Unable to give informed consent.
* Active hepatitis B (positive hepatitis B surface antigen (HBSAg) or HBSAg negative/ HB core antibody positive/ HBV PCR positive).
* Has substantial medical condition, that in the opinion of the investigator would preclude participation, as defined by

  * cardiovascular condition that may lead to an increased risk of complication if placed on study drugs.
  * gastrointestinal condition that would impair absorption of study drugs.
  * neurological or psychiatric condition that would significantly impair the ability to adhere to PrEP.
  * calculated GFR < 60 mL/min.
  * alcohol or drug abuse or dependence that would significantly impair the ability to adhere to PrEP (only for those with severe impairment).
  * other medical condition that would unacceptably increase the risk of harm from study drug or significantly impair the ability to adhere to PrEP.
* Suspected sensitivity or allergy to the study drug or any of its components.
* Currently using an essential product or medication that interacts with the study drug such as the following:

  * ART (including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents)
  * Agents with known nephrotoxic potential:

    * aminoglycoside antibiotics (including gentamicin)
    * IV amphotericin B
    * cidofovir
    * cisplatin
    * foscarnet
    * IV pentamidine
    * IV vancomycin
    * oral or IV gancyclovir
    * other agents with significant nephrotoxic potential
  * Drugs that slow renal excretion

    * Probenecid
  * Immune system modulators

    * Systemic chemotherapeutic agents (i.e. cancer treatment medications)
    * Ongoing systemic corticosteroids (with the exception of short courses of tapering steroid doses for asthma or other self- limited condition).
    * Interleukin-2 (IL-2)
    * Interferon (alpha, beta, or gamma)
  * Other agent known to have a significant interaction with TDF or FTC
  * Proteinuria 2+ or greater by urine dipstick
  * Signs or symptoms suggestive of acute HIV infection
  * Any other reason or condition that in the opinion of the investigator would interfere with participation, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Morris, MD, MPH, Principal Investigator — CCTG, UCSD AVRC; David Moore, PhD, Study Chair — CCTG, UCSD HNRP
Locations (4):
- United States (4):
  - City of Long Beach Department of Health and Human Services, Long Beach, California
  - University Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Pasipanodya EC, Jain S, Sun X, Blumenthal J, Ellorin E, Corado K, Dube MP, Daar ES, Morris SR, Moore DJ; California Collaborative Treatment Group (CCTG) TAPIR Study Team. Trajectories and Predictors of Longitudinal Preexposure Prophylaxis Adherence Among Men Who Have Sex With Men. J Infect Dis. 2018 Oct 5;218(10):1551-1559. doi: 10.1093/infdis/jiy368. PMID 30295803
- [Derived] Moore DJ, Jain S, Dube MP, Daar ES, Sun X, Young J, Corado K, Ellorin E, Milam J, Collins D, Blumenthal J, Best BM, Anderson P, Haubrich R, Morris SR. Randomized Controlled Trial of Daily Text Messages to Support Adherence to Preexposure Prophylaxis in Individuals at Risk for Human Immunodeficiency Virus: The TAPIR Study. Clin Infect Dis. 2018 May 2;66(10):1566-1572. doi: 10.1093/cid/cix1055. PMID 29228144

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SoC): Fixed-dose daily oral 300mg tenofovir (TDF) and 200mg emtricitabine (FTC) with Standard of Care (SOC)
- SoC + iTab: Fixed-dose daily oral 300mg tenofovir (TDF) and 200mg emtricitabine (FTC) with Standard of Care (SOC) and daily individualized text-messaging for adherence building (iTAB)
Period: Overall Study
Arm/Group | Standard of Care (SoC) | SoC + iTab
Started | 198 | 200
Completed | 166 | 158
Not Completed | 32 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | SoC + iTab | Total
Number analyzed (Participants) | 198 | 200 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.7) | 35.1 (9.8) | 35.2 (9.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 198 | 197 | 395
  Transgender woman | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 7 | 12
  Black | 26 | 26 | 52
  White | 148 | 147 | 295
  More than one race | 10 | 14 | 24
  Other | 4 | 3 | 7
  Hispanic ethnicity | 58 | 61 | 119
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 198 | 200 | 398
PREP use [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adherence to PrEP
Description: Proportion of participants adherent to PrEP as measured by TFV-DP dried blood spot (DBS) concentrations > 719 fmol/punch at Week 12 and the last on-drug visit.
Time Frame: Baseline to Week 48
Population: Only participants with a DBS sample collected at study visits were included in this analysis.
Measure: Number; unit: % participants with > 719 fmol/punch
Arm/Group | Standard of Care (SoC) | SoC + iTab
Number analyzed (Participants) | 181 | 180
% participants with > 719 fmol/punch
  Wk 12 | 85.6 | 91.7
  Wk 48 | 81.6 | 83.4

2. Secondary Outcome: Perfect Adherence to PrEP
Description: Proportion of participants with perfect adherence to PrEP as measured by TFV-DP dried blood spot (DBS) concentrations > 1246 fmol/punch at Week 12 and the last on-drug visit.
Time Frame: Baseline to Week 48
Population: Only participants with a DBS sample collected at study visits were included in this analysis.
Measure: Number; unit: % participants with > 1246 fmol/punch
Arm/Group | Standard of Care (SoC) | SoC + iTab
Number analyzed (Participants) | 181 | 180
% participants with > 1246 fmol/punch
  Wk 12 | 43.9 | 50.8
  Wk 48 | 37.4 | 51

3. Secondary Outcome: Rate of HIV Seroconversion
Description: Determine the rate of HIV seroconversion in PrEP users and compare the iTAB to SOC arms for number of new infections as a proportion at 48 weeks and end of study.
Time Frame: Up to 2.5 years after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | SoC + iTab
Number analyzed (Participants) | 198 | 200
Participants
  Wk 48 | 0 | 2
  End of Study | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to end of follow up for participants 0-120 weeks
Arm/Group | Standard of Care (SoC) | SoC + iTab
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/200
Serious Adverse Events (participants affected / at risk) | 1/198 | 2/200
Other Adverse Events (participants affected / at risk) | 15/198 | 21/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=198) | SoC + iTab (N=200)
Fanconi syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) — Related to study drug
HIV Seroconversion (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=198) | SoC + iTab (N=200)
GI symptoms (Gastrointestinal disorders) | 7 (8) | 12 (13) — nausea, diarrhea, abdomen pain
muscle pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
infection (Infections and infestations) | 1 (1) | 4 (4)
paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
depression with or without sucidality (Psychiatric disorders) | 2 (2) | 0 (0)
GU symptoms and disorders (Renal and urinary disorders) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
tonsil lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Discontinuation of PrEP may be for valid reasons for not needing prevention of HIV due to not being sexually active

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT01761643/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT01761643/SAP_001.pdf